

# Protocol for observational studies based on existing data

| <b>Document Number:</b> | c02336230-01 |
|---|---|
| BI Study No.: | 1160.207 |
| BI Investigational Product(s): | PRADAXA (dabigatran etexilate) |
| Title: | Sequential Expansion of Comparative Effectiveness of Oral<br>Anticoagulants: A Cohort Study |
| | (Phase 2 of the BI/ Pradaxa study program) |
| Title for lay people: | Comparative effectiveness of oral anticoagulants |
| Date of last version of protocol: | 25 Feb 2014 |
| EU PAS Register No:<br>only applicable for PASS | N/A |
| Marketing authorization holder(s): | Boehringer Ingelheim |
| Author / Responsible<br>Parties/BI contact<br>person: | . All from the |
| Country(-ies) of study: | US |
| Status: | Final Protocol |
| EU-QPPV: only applicable for PASS | |
| Signature of EU-QPPV:<br>only applicable for PASS | |
| Version and Date: | Version 1, 25 Feb 2014 |

**Proprietary confidential information** 

© 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## PROTOCOL ABSTRACT

| Name of company: | | | O P 1 : |
|---|---|---|---|
| Boehringer Ingelheim | | | Boehringer Ingelheim |
| Name of product: | Name of product: | | |
| PRADAXA <sup>®</sup> | | | |
| Name of active ingredie<br>DABIGATRAN ETEXIL | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 25 Feb 2014 | 1160.207 | Version 1 | 25 Feb 2014 |
| | lheim International GmbH | confidential information I or one or more of its affiliated compreproduced, published or otherwise used with | |
| Title of study: | Sequential expansion of study | f comparative effectiveness of oral a | anticoagulants: a cohort |
| Team member<br>Epidemiology: | | | |
| Project team: | | | |
| Rationale and background: | A number of new oral anticoagulants are being developed and marketed to replace vitamin K antagonists. Unlike vitamin K antagonists, these new drugs do not require dose titration involving intensive therapeutic monitoring of prothrombin time to achieve target anticoagulation within a narrow therapeutic range. However, their long-term safety and effectiveness have not been characterized in a real-world setting. | | |
| Research question and objectives: | This protocol is for a series of comparative effectiveness and safety analyses within periodically updated cohorts of patients initiating dabigatran (compared to warfarin) and other new oral anticoagulants (NOAC) (as they become available), compared to warfarin, followed longitudinally for the occurrence of a variety of health outcomes. | | |
| | <ol> <li>Objectives</li> <li>Primarily, to conduct direct comparisons over time between dabigatran and warfarin and quantify the association between anticoagulant choice and the occurrence of specific outcomes of interest</li> <li>Secondarily, to monitor the number of people initiating other NOAC medications and, when sufficient, to compare study outcomes between other NOAC medications and warfarin</li> </ol> | | |
| Study design: | Observational sequent | ial cohort study based on existin | g data |

| Name of company: | | | Boehringer |
|---|---|---|---|
| Boehringer Ingelheim | | | Ingelheim |
| Name of product: | | | |
| PRADAXA <sup>®</sup> | | | |
| Name of active ingrediction DABIGATRAN ETEX | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 25 Feb 2014 | 1160.207 | Version 1 | 25 Feb 2014 |
| | elheim International GmbH<br>in full or in part - be passed on, 1 | confidential information I or one or more of its affiliated compreproduced, published or otherwise used with a diagnosis of atrial fibrillation | hout prior written permission |
| 1 opulation. | Patients with a recorded diagnosis of atrial fibrillation without evidence of valvular etiology who initiate dabigatran (or other NOACs as they become available) compared with warfarin initiators. | | |
| Study data source: | This study will be conducted within both UnitedHealth and Marketscan data sources. The first analyses of this study will include data from October 2010 through December 2012 for the cohort formation and data from July 2008 through September 2010 for disease risk score (DRS) calculation. Both data sources will be updated on a 6-month basis through December 2015 | | |
| Expected study size: | Sources will be updated on a 6-month basis through December 2015 The estimated final study size will be ~ 60,000 dabigatran initiators, matched to ~60,000 warfarin initiators with approximately 24,000 cumulative personyears of observation in each exposure group, and other NOAC initiators (numbers dependent on use) separately matched to a similar number of warfarin initiators. The estimated study size (after PS matching) for interim analyses: Interim report 1 (Apr 2014): ~ 24,000 dabigatran and ~24,000 warfarin initiators with 10,000 PYs of observation in each group Interim report 2 (Jul 2014): ~ 30,000 dabigatran and ~30,000 warfarin initiators with 12,350 PYs of observation in each group Interim report 3 (Nov 2014): ~ 36,000 dabigatran and ~36,000 warfarin initiators with 14,700 PYs of observation in each group Interim report 4 (Mar 2015): ~ 42,000 dabigatran and ~42,000 warfarin initiators with 17,050 PYs of observation in each group Interim report 5 (Sep 2015): ~ 48,000 dabigatran and ~48,000 warfarin initiators with 19,400 PYs of observation in each group Interim report 6 (Mar 2016): ~ 54,000 dabigatran and ~54,000 warfarin initiators with 21,750 PYs of observation in each group Final report (Dec 2016): ~ 60,000 dabigatran and ~60,000 warfarin initiators with 24.100 PYs of observation in each group | | |

| Name of company: | | | Boehringer |
|---|---|---|---|
| Boehringer Ingelheim | | | Ingelheim |
| Name of product: | | | |
| PRADAXA <sup>®</sup> | | | |
| Name of active ingredi<br>DABIGATRAN ETEXI | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 25 Feb 2014 | 1160.207 | Version 1 | 25 Feb 2014 |
| © 2014 Boehringer Ing This document may not - Main criteria for inclusion: | Proprietary confidential information CHA2DS2-VASc score ≥ 1 International Graph or one or more of its affiliated companies. All rights reserved. | | |
| Main criteria for exclusion: | <ul> <li>Patients with missing or ambiguous age or sex information.</li> <li>Patients with evidence of valvular disease.</li> <li>Patients with less than 12 months enrolment preceding the date of anticoagulant initiation</li> <li>Patients with a dispensing of any oral anticoagulant during the 12 months preceding the date of anticoagulant initiation</li> <li>Patients with a nursing home stay during baseline</li> </ul> | | |
| Comparison group: | Warfarin | | |
| Expected duration of exposure: | As observed in the data source | | |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## TABLE OF CONTENTS

| TITLE | PAGE | 1 |
|--------------|-------------------------------------------------|----|
| PROTO | OCOL ABSTRACT | 2 |
| TABLE | OF CONTENTS | 5 |
| LIST O | OF TABLES | 7 |
| | F FIGURES | |
| 1. | LIST OF ABBREVIATIONS AND TERMS | |
| 2. | RESPONSIBLE PARTIES | |
| 3. | AMENDMENT AND UPDATES | |
| 4. | MILESTONES | |
| 5. | RATIONALE AND BACKGROUND | 14 |
| 6. | RESEARCH QUESTIONS AND OBJECTIVES | 15 |
| <b>7.</b> | RESEARCH METHODS | 16 |
| 7.1 | STUDY DESIGN | 16 |
| 7.2 | SETTING | |
| 7.3 | SUBJECTS | 17 |
| 7.4 | VARIABLES | 19 |
| <b>7.4.1</b> | EXPOSURES | 19 |
| 7.4.2 | OUTCOME(S) | 21 |
| 7.5 | DATA SOURCES | 36 |
| <b>7.6</b> | BIAS | 37 |
| 7.7 | STUDY SIZE | |
| 7.9 | DATA ANALYSIS | 40 |
| 7.9.1 | MAIN ANALYSIS | |
| 7.10 | QUALITY CONTROL | 15 |
| 7.10<br>7.11 | LIMITATIONS OF THE RESEARCH METHODS | |
| 7.12 | OTHER ASPECTS | |
| 8. | PROTECTION OF HUMAN SUBJECTS | 47 |
| 9. | MANAGEMENT AND REPORTING OF ADVERSE | |
| | EVENTS/ADVERSE REACTIONS | 48 |
| 10. | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY | |
| | RESULTS | 49 |
| 11. | REFERENCES | 50 |
| 12. | FUNDING | 53 |

| Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companie |
|---|

| 13. | ANNEX | 54 |
|-------|----------------------------------|----|
| ANNEX | 1: LIST OF STAND-ALONE DOCUMENTS | 54 |
| ANNEX | 3 EXAMPLE STUDY SHELL TABLES | 65 |
| ANNEX | 4 STUDY FIGURES | 73 |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## LIST OF TABLES

| Table 1<br>Table 2 | Market availability for the treatments of interest. Outcome Definitions. | |
|---|---|---|
| Table 7 | UnitedHealth and MarketScan databases, estimated numbers of dabigatran and warfarin with non-valvular atrial fibrillation diagnosis, | |
| | in the period October 2010 – June 2012 | 37 |
| Table 8 | Projected minimum detectable relative rates* by reporting period | 38 |
| Table A3 | Follow-up and outcomes among matched cohorts | 70 |
| Table A4 | Follow-up and distribution of reasons for discontinuation | 71 |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## LIST OF FIGURES

| Figure 1 | Patient Selection Flow | 19 |
|-----------|------------------------------------------------|----|
| Figure A1 | Patient Selection Flow Diagram (CONSORT Style) | 73 |
| Figure A2 | Survival curves (time to event) | 74 |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. LIST OF ABBREVIATIONS AND TERMS

ACCP American College of Chest Physicians
ACEI Angiotensin-converting Enzyme Inhibitor

AES Advanced Encryption Standard

AF Atrial Fibrillation

ALT Serum Alanine Aminotransferase ARB Angiotensin Receptor Blocker

ASCVD Atherosclerotic Cardiovascular Disease

BB Beta Blocker

BI Boehringer Ingelheim BMI Body Mass Index

CABG Coronary Artery Bypass Graft
CAD Coronary Artery Disease
CCB Calcium Channel Blocker

CHA<sub>2</sub>DS<sub>2</sub>-VASc Congestive Heart Failure, Hypertension, Age > 75, Diabetes

Mellitus, Prior Stroke or Transient Ischemic Attack, Vascular

Disease, Age 65-74, Sex Category

CHADS<sub>2</sub> Congestive Heart Failure, Hypertension, Age> 75, Diabetes

Mellitus, Prior Stroke or Transient Ischemic Attack

CHF Congestive Heart Failure
CI Confidence Interval

CONSORT Consolidated Standards for Reporting Trials

CPT Current Procedural Terminology

Cr Creatinine

DM Diabetes Mellitus

DRG Disease

DRS Disease Risk Score

DVT Deep Venous Thromboembolism

Dx Diagnosis-Related Group

ESC European Society of Cardiology
GFR Glomerular Filtration Rate

GI Gastrointestinal

H2 Receptor Histamine H2 Receptor

HAS-BLED Hypertension, Abnormal Liver/Renal function, Stroke, Bleeding

history or predisposition, Labile INR, Elderly (Age >65), Drugs-

Alcohol usage

HbA1c Hemoglobin A1C

HCPC Healthcare Common Procedure Coding hdPS High-dimensional Propensity Score

HR Hazard Ratio

ICD-9 International Classification of Diseases, Ninth Revision, Clinical

Modification

### Boehringer Ingelheim Protocol for observational studies based on existing data


**1160.207** c02336230-01

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

ICH Intracerebral Hemorrhage INR International Normalized Ratio

ITT Intent-To-Treat

LDL Low Density Lipoprotein

LOS Length of Stay

MDRD Modification of Diet in Renal Disease

MI Myocardial Infarction NOAC New Oral Anticoagulant

NSAID Non-steroidal Anti-inflammatory Drug

NVAF Non-valvular Atrial Fibrillation PAD Peripheral Artery Disease

PCI Percutaneous Coronary Intervention

PE Pulmonary Embolism

PGP P-glycoprotein

PPI Proton Pump Inhibitor
PPV Positive Predictive Value

PS Propensity Score

PTCA Percutaneous Transluminal Coronary Angioplasty

PVD Peripheral Vascular Disease

PY Person-Year

RE-LY Randomized Evaluation of Long-Term Anticoagulation Therapy

RR Relative Risk

SAH Subarachnoid Hemorrhage

SCr Serum Creatinine SD Standard Deviation

TIA Transient Ischemic Attack

US United States

VTE Venous Thromboembolism

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. RESPONSIBLE PARTIES

(1) (1) (1) (1)

(1)

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. AMENDMENT AND UPDATES

None

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. MILESTONES

Planned dates for the following milestones:

| Date | Phase 2 | | Data Source | |
|---|---|---|---|---|
| | Milestone | Month | United | MarketScan |
| | | | Claims and lab data are released<br>every 6 months in Jan and Jul<br>(6-month lag time) | Claims data are released quarterly in Mar, Jun, Sept, and Dec (9-month lag time) Lab data are released yearly in Dec (12-month lag time) |
| Jun, 2012 | Contract | 0 | | |
| | Year 1 | 1 | | |
| Jun, 2013 | Draft Protocol | 12 | | |
| | | _ | Year 2 | |
| Jan, 2014 | Final Protocol | 19 | | |
| Apr, 2014 | Interim Report 1 | 22 | Data through Dec 2012 | Claims through Dec 2012 Labs through Dec 2012 |
| Jul, 2014 | Interim Report 2 | 25 | Data through Jun 2013<br>(Update received in Jan 2014) | Claims through Jun 2013 (Update received in Mar 2014) Labs through Dec 2012 (Update received in Dec 2013) |
| Nov, 2014 | Interim Report 3 | 29 | Data through Dec 2013<br>(Update received in Jul 2014) | Claims through Sep 2013 (Update received in Jun 2014) Labs through Dec 2012 (Update received in Dec 2013) |
| | Year 3 | | | |
| Mar, 2015 | Interim Report 4 | 32 | Data through Jun 2014<br>(Update received in Jan 2015) | Claims through Dec 2013 (Update received in Dec 2014) Labs through Dec 2013 (Update received in Dec 2014) |
| Sep, 2015 | Interim Report 5 | 39 | Data through Dec 2014<br>(Update received in Jul 2015) | Claims through Sep 2014 (Update received in Jun 2015) Labs through Dec 2013 (Update received in Dec 2014) |
| | T | _ | <u>Year 4</u> | |
| Mar, 2016 | Interim Report 6 | 45 | <u>Data through Jun 2015</u><br>(Update received in Jan 2016) | Claims through Dec 2014 (Update received in Dec 2015) Labs through Dec 2014 (Update received in Dec 2015) |
| | Year 4 | <b>-</b> | | |
| Dec, 2016 | Final Report | 54 | <u>Data through Dec 2015</u><br>(Update received in Jul 2016) | Claims through Dec 2015 (Update received in Sep 2016) Labs through Dec 2014 (Update received in Dec 2054) |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. RATIONALE AND BACKGROUND

A number of new oral anticoagulants are being developed and marketed to replace vitamin K antagonists, one of the most important drugs in modern medicine. [P11-11875] Unlike vitamin K antagonists, these new drugs do not require dose titration involving intensive therapeutic monitoring of prothrombin time to achieve target anticoagulation within a narrow therapeutic range. In Phase III studies, these drugs were found to be therapeutically advantageous or non-inferior over warfarin. In the coming years, as many as six new anticoagulants could be on the market and a lack of valid comparative evidence will hinder prescriber and payor decision-making.

To date, these drugs have been studied in randomized clinical trials for three separate indications: (1) prevention of stroke and systemic embolism among patients with atrial fibrillation; (2) prevention of deep venous thrombosis (DVT) among patients undergoing hip or knee replacement therapy; and (3) treatment of venous thromboembolism (VTE). Phase III clinical trials comparing dabigatran, rivaroxaban, apixaban, and edoxaban to warfarin in patients with non-valvular atrial fibrillation (NVAF) have been completed. [R11-4190] [P09-11669] [R11-4223] [R13-5082] The objective of this part of the project is to conduct a series of comparative effectiveness and safety studies across the available anticoagulants, starting with warfarin and dabigatran and including additional ones as they become available within data sources available to us at the Division of Pharmacoepidemiology. Such sequential approach will extend Phase I analyses (study protocol 1160.157) by providing greater precision around effect estimates as well as providing an evaluation of their use in actual practice and among subgroups of patients that were not represented in clinical trials. This evaluation will provide a direct assessment of comparative effectiveness and potential adverse events across the anticoagulants that may have eluded the pre-marketing trials.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. RESEARCH QUESTIONS AND OBJECTIVES

This protocol is for a series of comparative effectiveness and safety analyses within periodically updated cohorts of patients with NVAF at risk for stroke initiating dabigatran or other oral NOAC medications as they become available, compared to warfarin, followed longitudinally for the occurrence of a variety of health outcomes.

Specific objectives of this active surveillance program are:

- 1) Primarily, to conduct direct comparisons over time between dabigatran and warfarin and quantify the association between anticoagulant choice and the occurrence of specific outcomes of interest
- 2) Secondarily, to monitor the number of people initiating other NOAC medications as they become available and, when sufficient, to compare study outcomes between other NOAC medications and warfarin.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RESEARCH METHODS

#### 7.1 STUDY DESIGN

This study will involve a sequentially built parallel cohort design with propensity score (PS) matching to address potential confounding. Each new data update will provide additional follow-up time on the patients already in the cohort, as well as new initiators who will be matched on PS and calendar quarter of initiation and added to the existing cohort for the cumulative analyses. This study design was selected to facilitate the inclusion of additional subjects and follow-up time as data become available over the course of the study period. The study will be conducted within two US-based longitudinal healthcare claims databases (MarketScan and UnitedHealth Research Database, see also section 6.5 for more details). Cohort selection and all analyses will be performed separately within each database and a combined analysis that pools results from the two databases for the same time periods will be done if appropriate, based on an assessment of homogeneity of treatment effect. Pooling of results across data sources will correspond to a weighted average effect (as in a fixed effects meta-analysis) using the Mantel-Haenszel method. [R97-0509] It is expected that there will be little heterogeneity of treatment effects across the databases since the databases are similar with respect to who is included in the database (employed people and their dependents) and the nature of data captured (health insurance transactions billed on a negotiated fee for service basis). Heterogeneity will be assessed by comparing the treatment effect point estimates across data sources. Assessment of heterogeneity will not rely on a statistical test of heterogeneity, since the large study size may indicate significant heterogeneity (p<0.05) even if estimates are similar (i.e. a difference that is not clinically meaningful) and the purpose of this assessment of heterogeneity is intended only for determining whether it is reasonable to combine data sources. If contrary to expectations, there is a difference >30% in the overall effect measure for a primary outcome across the two data sources, we will conduct an additional investigation that assesses treatment effect within levels of protocol-specified subgroups (Section 6.9.2) separately by a database. If treatment effect is different across levels of the subgroup variable within a data source, and the distribution of this subgroup variable differs by data source, then the pooling will be conducted within strata of the subgroup variable or variables across which heterogeneity is observed to account for this heterogeneity.

The primary analyses will involve dabigatran initiators compared to warfarin initiators; as other NOAC medications become available for stroke prevention, we will form additional cohorts of other NOAC medications and separately compare them to warfarin in the secondary analyses once sufficient number of initiators will have accrued. The same (as described below for dabigatran) inclusion/exclusion criteria will apply and a similar set of analyses will be conducted.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.2 SETTING

Initiators of dabigatran and warfarin from two US data sources: (1) UnitedHealth Research Database and (2) MarketScan Commercial Claims and Encounters database and Medicare supplement between October 2010 and December 2012, with 6-month updates through December 2015. Initiators of other NOAC medications will be added as these medications become available for stroke prevention in NVAF. Data from July 2008 through September 2010 will be used for disease risk score (DRS) calculation.

#### 7.3 SUBJECTS

#### Patient Selection:

- The main cohort will consist of patients with NVAF at risk for stroke initiating an oral anticoagulant medication in the timeframe of the study
  - warfarin and dabigatran for the primary analysis
  - other NOACs to be added separately in the secondary analysis as they become available for stroke prevention in later time intervals
- Warfarin initiators between January 2009 and September 2010 will be used for estimation of disease risk scores.

#### Inclusion criteria:

- Initiation of an oral anticoagulant is defined by a dispensing of an anticoagulant medication (warfarin or a NOAC medication) in the source data, with no dispensing of any oral anticoagulant in the prior 12 months. The date of that dispensing will be defined as the index date for that initiation.
- At least one ICD-9 diagnosis code of 427.31 (atrial fibrillation) at any time prior to and including the index date
- At least 12 months (365 days) continuous enrollment, defined as ≤32 days enrollment gap using enrollment and disenrollment dates, preceding the index date
- 18 years of age and older at index date
- $CHA_2DS_2$ -VASc score  $\geq 1$

#### Exclusion criteria:

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Patients with missing or ambiguous age or sex information
- Patients with a nursing home stay during baseline
- Patients with a dispensing of any oral anticoagulant during the 12 months preceding and including the index date
- Patients with documented evidence of valvular disease defined as at least 1 inpatient or outpatient ICD-9 Dx code of [R11-4334]

394.x (diseases of mitral valve)

395.x (diseases of aortic valve)

396.x (diseases of mitral and aortic valve)

397.x (diseases of other endocardial structures)

398.9x (other and unspecified rheumatic heart diseases)

V42.2 (heart valve replaced by transplant)

V43.3 (heart valve replaced by a mechanical device/prosthesis)

OR

ICD-9 procedure code 35.1x (open heart valvuloplasty without replacement), 35.2x (replacement of heart valve) [R03-1232]

OR

one of the following CPT codes:

33660-33665 (atrioventricular valve repair)

33400-33403 (aortic valve valvuloplasty)

33420-33430 (mitral valve repair/valvuloplasty/replacement)

33460 (valvectomy, tricuspid valve, with cardiopulmonary bypass)

33463-33468 (tricuspid valve repair/valvuloplasty/replacement)

33475 (replacement, pulmonary valve)

33496 (prosthetic valve dysfunction repair)

0257T (implantation of catheter-delivered prosthetic aortic heart valve; open thoracic approach)

0258T (transthoracic cardiac exposure for catheter-delivered aortic valve replacement; without cardiopulmonary bypass)

0259T (transthoracic cardiac exposure for catheter-delivered aortic valve replacement; with cardiopulmonary bypass)

0262T (implantation of catheter-delivered prosthetic pulmonary valve, endovascular approach)

at any time prior to and including the index date.

We will balance baseline covariates among patients initiating each drug by means of a multivariate confounder summary score (by matching on the exposure propensity score, with confounder balance assessed by the disease risk score). [R12-1912]

#### Cohort formation

We will receive new data as they become available on a periodic basis (every 6 months) and we will update the study cohorts through December 2015. Initiators of oral anticoagulants identified in each data cut, as previously described, will form sequential cohorts.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In each sequential cohort we will balance baseline covariates among patients initiating each drug by matching on the exposure propensity score and calendar quarter of initiation. Patients' follow-up will end when there is a treatment gap of  $\geq 14$  days from the end of calculated days supplied. Patients will be allowed to contribute only once.



Figure 1 Patient Selection Flow

#### 7.4 VARIABLES

#### 7.4.1 EXPOSURES

Table 1 Market availability for the treatments of interest

| Class | Drug | FDA approved* | FDA approved for stroke prevention ir<br>patients with non-valvular atrial<br>fibrillation at risk for stroke |
|---|---|---|---|
| Direct<br>thrombin<br>inhibitors | <br>Dabigatran | 19 October 2010 | 19 October 2010 |
| Direct Xa | Rivaroxaban | 1 July 2011 | 4 November 2011 |
| inhibitors | Apixaban | 28 December 2012 | 28 December 2012 |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Table 1 (con't) Market availability for the treatments of interest

| Edoxaban | Phase III | N/A |
|------------|-----------|-----|
| Otamixaban | Phase III | N/A |
| Betrixaban | Phase II | N/A |

<sup>\*</sup>as of December 2013

The primary contrast of interest is between new initiators of warfarin and new initiators of dabigatran, defined as no anticoagulation with *any oral anticoagulant* in the 12 months before the index prescription.

In the secondary analysis and as they become available for stroke prevention in NVAF patients, other NOAC medications will be compared to warfarin. The same definitions and inclusion/exclusion criteria will be applied.

Concomitant therapy with medications that are not cohort-defining medications (defined as simultaneous use on the day of dabigatran or warfarin initiation) will be accounted for in the study analyses as a covariate and used for balancing or stratification.

### Study follow-up

We will follow patients for each of the outcomes of interest in a prospective manner and we will estimate measures of effect using person-time based analyses.

The primary analyses will use an 'as treated' approach. Follow-up will start the day after cohort inclusion, which is the day of treatment initiation, and will end at the time of disenrollment, end of the observation period (available data), death, admission to a nursing home, discontinuation of the index study exposure, or switch to a different anticoagulant whichever comes first. Exposure will be considered discontinued if there is a treatment gap ≥14 days from the end of calculated days supplied. Warfarin therapy involves dose titration following initiation before a stable therapeutic INR is obtained. We will use the reported days' supply as a proxy for duration of exposure following a dispensing as it may more adequately reflect the use pattern within a commercial health insurer database represented by UnitedHealth and MarketScan. This approach involves a potential mismatch between the presumed exposure derived from dispensing data and actual exposure. The utilization study (described in study protocol 1160.177) will inform the sensitivity analyses around this assumption and seek to clarify how sensitive results are to variations in the exposure assumption. Switchers will be censored in the as-treated approach on the day of the dispensing of the alternative medication. If switching was the consequence of a side effect of a drug, most likely the index drug was discontinued for some time before the new drug was initiated. Any clinical event therefore was most likely recorded during that period and will be

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

attributed to the index drug.

#### 7.4.2 **OUTCOME(S)**

The primary outcomes of interest include stroke (hemorrhagic, ischemic, uncertain classification) and major bleeding. Secondary outcomes are: stroke or systemic embolism, transient ischemic attack (TIA), myocardial infarction (MI), venous thromboembolism (VTE), deep vein thrombosis (DVT), pulmonary embolism (PE). Systemic embolism (defined as an acute vascular occlusion of the extremities or any organ.

Systemic embolism (defined as an acute vascular occlusion of the extremities or any organ, such as kidneys, mesenteric arteries, spleen, retina or grafts), ischemic stroke, hemorrhagic stroke, stroke of uncertain classifications, major intracranial bleeding, major extracranial bleeding, major gastrointestinal (GI) bleeding, major upper GI bleeding, major lower GI bleeding, major urogenital bleeding, major other bleeding. Further outcomes include hepatotoxicity and all-cause mortality.

As mortality data in the commercial databases is currently limited to inpatient deaths, we will seek to improve the ascertainment of the death outcome through external linkage, such as with the Social Security Death Master File.

Table 2Outcome Definitions

| Outcome | Hospital Discharge Code(s) | Comments |
|---|---|---|
| Primary Outcome | Primary Outcomes | |
| Stroke | <u> </u> | See Mini-Sentinel report |
| | 431.x Intracerebral hemorrhage (ICH) | for PPV for individual |
| | 433.x1 Occlusion and stenosis of precerebral arteries with | codes or other algorithms |
| | cerebral infarction | [ <u>R14-0052</u> ] |
| | 434.x1 Occlusion and stenosis of cerebral arteries with | |
| | cerebral infarction | |
| | 436.x Acute, but ill-defined cerebrovascular events | |
| Major | Major intracranial bleeding, major extracranial bleed | |
| hemorrhage | (for codes see component outcomes below) | |
| Secondary outcomes | | |
| Stroke or | Stroke or systemic embolism (for codes see component | |
| systemic | outcomes below) | |
| embolism | | |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Table 2 (con't) Outcome Definitions

| Outcome | Hospital Discharge Code(s) | Comments |
|----------|----------------------------|------------------------|
| Systemic | ICD-9 Diagnoses: | No validation studies |
| embolism | 444.x Arterial embolism | available. Codes are |
| | | thought to be specific |
| | | because of the |
| | | substantial clinical |
| | | symptomatic and |
| | | required therapy. |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Table 2 (con't) Outcome Definitions

| Ischemic stroke | As primary ICD-9 discharge diagnosis (Dx): ICD-9 Dx 433.x1 Occlusion and stenosis of precerebral | PPV 95.5% in commercially-insured |
|---|---|---|
| | arteries with cerebral infarction | population for the |
| | ICD-9 Dx 434.x1 Occlusion and stenosis of cerebral | codes in any position |
| | arteries with cerebral infarction | [ <u>R11-4887</u> ] |
| | | Use of codes in the |
| | | primary position |
| | | generally increases the |
| | | PPVs [ <u>R14-0052</u> ] |
| Hemorrhagic | As primary ICD-9 discharge diagnosis (Dx): | Median PPV 96% |
| stroke | 431.x Intracerebral hemorrhage (ICH) | (86% if all discharge |
| | | diagnoses) for ICH |
| | | based on 2 validation |
| | | studies [ <u>R14-0052</u> ] |
| Stroke | As primary ICD-9 discharge diagnosis (Dx): | Mini-Sentinel report: |
| uncertain | ICD-9 Dx code 436.x (acute, but ill-defined | Median PPV of 81% |
| classification | cerebrovascular disease) | for the code of 436 |
| | | [R14-0052] |
| Transient | ICD-9 Dx code 435.xx (transient cerebral ischemia) as | PPV of 89% (primary |
| Ischemic | the principal (primary) discharge diagnosis | Dx) and 77% (primary |
| Attack (TIA) | | and secondary) in 1992 |
| , , | | study [R13-0519] and |
| | | 70% (primary only in |
| | | Canadian database) |
| | | [ <u>R13-0520</u> ] have been |
| | | reported. |
| | | Median PPV is 79% |
| | | (72 if all discharge Dx) |
| | | [ <u>R14-0052</u> ] |
| Myocardial | ICD-9 Dx 410.X (acute myocardial infarction) | PPV 94% in Medicare |
| infarction (MI) | excluding 410.x2 (subsequent episode of care), as the | claims data [ <u>R11-4316</u> ] |
| | principal (primary) or the next (secondary) diagnosis | PPV 88.4% in |
| | AND | commercially-insured |
| | a length of stay (LOS) between 3-180 days, or death if | population [ <u>R11-4887</u> ] |
| | LOS is < 3 days | |
| Venous | DVT or PE (for codes see component outcomes below) | |
| Thromboembol | | |
| ism (VTE) | | |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **Table 2 (con't) Outcome Definitions**

| Door vein | Validated algorithms | Algorithm for Door |
|---|---|---|
| Deep vein | Validated algorithm: | Algorithm for Deep |
| thrombosis | ICD-9 451.1x (Phlebitis and thrombophlebitis of deep | vein thrombosis |
| (DVT) | vessels of lower extremities) | (DVT): ICD-9 codes of |
| | ICD-9 451.2x (of lower extremities, unspecified) | 451.1, 451.2, 451.81, |
| | ICD-9 451.81 (of Iliac vein) | 451.9, 453.1, 453.2, |
| | ICD-9 451.9x (of unspecified site) | 453.8, 453.9 [hospital |
| | ICD-9 453.1x (thrombophlebitis migrans) | discharge, any |
| | ICD-9 453.2x (venous embolism and thrombosis of | position] had PPV of |
| | vena cava) | 0.72 and specificity > |
| | ICD-9 453.8x (venous embolism and thrombosis of | 0.99 in Medicare |
| | other specified veins) | population [ <u>R11-4334</u> ] |
| | ICD-9 453.9x (venous embolism and thrombosis of | |
| | unspecified site) | |
| | Not in the validated algorithm but will be included | Mini-Sentinel: while |
| | following Mini-Sentinel recommendation for VTE | using ICD-9 codes |
| | outcome: | 415.x (PE), 451.x and |
| | ICD-9 453.40 (Venous embolism and thrombosis of | 453.x (DVT) as a VTE |
| | unspecified deep vessels of lower extremity (includes | event yielded the |
| | DVT) | highest PPV, for a |
| | ICD-9 453.41 (Venous embolism and thrombosis of | specific event (DVT or |
| | deep vessels of proximal lower extremity (includes | PE) PPV was lower; |
| | femoral, iliac, popliteal, thigh, and upper leg) | therefore, the |
| | ICD-9 453.42 (Venous embolism and thrombosis of | performance of |
| | deep vessels of distal lower extremity (includes calf, | algorithms depends on |
| | lower leg, peroneal, and tibia) | a population studied |
| | ICD-9 453.0 (Hepatic vein thrombosis) | [ <u>R13-0522</u> ] |
| Pulmonary | ICD-9 415.1x (pulmonary embolism and infarction) | PPV of 72% in a |
| Embolism (PE) | Teb y 1701711 (paintenary time enoisin and interestion) | community sample (45 |
| Emoonsm (1 L) | | YO and older) [R05- |
| | | 0358] |
| Major | ICD-9 diagnosis: | PPV 77% or higher |
| intracranial | 430.x (Subarachnoid hemorrhage (SAH)) | reported [ <u>R14-0052</u> ] |
| bleeding | 431.x (Intracerebral hemorrhage (ICH)) | [ <u>K14-0032</u> ] |
| biccamg | 432.x (other and unspecified intracranial hemorrhage, | |
| | including 432.1x – subdural hemorrhage) | |
| Major | Major upper GI bleed, major lower and unspecified GI | No validation studies |
| extracranial | bleed, major urogenital bleed, major other bleed (for codes | available for this |
| bleeding | | |
| | see component outcomes below) | outcome |
| Major GI | Major upper GI bleeding, major lower/unspecified GI | No validation studies |
| bleeding | bleeding (for codes see component outcomes below) | available for this |
| | | outcome |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **Table 2 (con't) Outcome Definitions**

| Major upper | ICD-9 diagnoses: | PPV of 87.8% in |
|---|---|---|
| GI bleed | 531.0x (acute gastric ulcer with hemorrhage with/without | commercially-insured |
| Of bleed | obstruction) | population [R11-4887] |
| | 531.2x (with hemorrhage and perforation with/without | population [ <u>K11-4887</u> ] |
| | obstruction) | |
| | 531.4x (chronic or unspecified gastric ulcer with hemorrhage | |
| | with/without obstruction) | |
| | 531.6x (with hemorrhage and perforation with/without | |
| | obstruction) | |
| | 532.0x (acute duodenal ulcer with hemorrhage with/without | |
| | obstruction) | |
| | 532.2x (with hemorrhage and perforation with/without | |
| | obstruction) | |
| | 532.4x (chronic or unspecified duodenal ulcer with | |
| | hemorrhage with/without obstruction) | |
| | 532.6x (with hemorrhage and perforation with/without | |
| | obstruction) | |
| | 533.0x (acute peptic ulcer of unspecified site with | |
| | hemorrhage with/without obstruction) | |
| | 533.2x (with hemorrhage and perforation with/without obstruction) | |
| | 533.4x (chronic or unspecified peptic ulcer of unspecified site | |
| | with hemorrhage with/without obstruction) | |
| | 533.6x (with hemorrhage and perforation with/without | |
| | obstruction), | |
| | 534.0x (acute gastrojejunal ulcer with hemorrhage | |
| | with/without obstruction) | |
| | 534.2x (with hemorrhage and perforation with/without | |
| | obstruction) | |
| | 534.4x (chronic or unspecified gastrojejunal ulcer with | |
| | hemorrhage with/without obstruction) | |
| | 534.6x (with hemorrhage and perforation with/without | |
| | obstruction) | |
| | 578.0 (hematemesis) OR | |
| | ICD-9 procedure code 44.43 (endoscopic control of gastric or | |
| | duodenal bleeding) OR | |
| | CPT code 43255 (upper gastrointestinal endoscopy including | |
| | esophagus, stomach, and either the duodenum and/or jejunum as appropriate with control of bleeding, any method) | |
| Major lower | Lower GI/unspecified GI site bleeds [R11-2274]: | PPVs for individual |
| GI bleeding | Diverticulosis of small intestine with hemorrhage: | codes [ <u>R11-2274</u> ]: |
| Of bleeding | 562.02 | 562.12 - 91.7% |
| | | 562.13 – 66.7% |
| | Diverticulitis of small intestine with hemorrhage: | 569.3 - 71.4% |
| | 562.03 Diverticularie of colon with homeomhogo, 562.12 | |
| | Diverticulosis of colon with hemorrhage: 562.12 | 569.85 – 100% |
| | Diverticulitis of colon with hemorrhage: 562.13 | 578.1 - 81.8% |
| | Hemorrhage of rectum and anus: 569.3x | 578.9 -88.2% |
| | Angiodysplasia of intestine with hemorrhage: 569.85 | |
| | Blood in stool: 578.1x | |
| | Hemorrhage of GI tract, unspecified: 578.9 | |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Table 2 (con't) Outcome Definitions

| Major<br>urogenital<br>bleed | ICD-9 diagnoses: Hematuria: ICD-9 Dx: 599.7 Excessive/frequent menstruation: ICD-9 Dx 626.2x and secondary diagnosis indicating acute bleeding: anemia (280.0, 285.1, 285.9), [R11-2274] | PPVs for individual codes [R11-2274]: 599.7 - 75.0% 626.2 - 100% (2 cases) [R11-2274] |
|---|---|---|
| Other major bleeds | Other major bleeds [R11-2274]: Hemathrosis: 719.1x Hemopericardium: 423.0x Hemoptysis: 786.3x Epistaxis: 784.7x Hemorrhage not specified 459.0x Acute posthemorrhagic anemia 285.1x | PPVs for individual codes [R11-2274]: 719.1x - 100% 786.3x - 80% 784.7x - 100% 459.0x - 100% 285.1x - 100% |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.5 DATA SOURCES

The data source for this project will be a combination of claims data from United Healthcare, a large national commercial health insurer, and MarketScan, a research claims database from commercial employer-sponsored health plans from July 2008 through December 2012 for the first interim report, with 6-month updates through December 2015. Data from July 2008 through September 2010 will be used for DRS estimation (see Main Analysis Section (6.9.1) for more details) while data from October 2010 will be used for cohort formation and analysis. Because of a 6-month time lag before data become available for United and 9-month time lag for MarketScan, we will not have access to any information beyond December 2012 for the first interim report.
Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

•

We have obtained the following preliminary estimates from the UnitedHealth and MarketScan databases regarding the number of patients initiating dabigatran or warfarin (new users) and meeting the main study selection criteria in the period October 2010 – June 2012.

Table 7 UnitedHealth and MarketScan databases, estimated numbers of dabigatran and warfarin with non-valvular atrial fibrillation diagnosis, in the period October 2010 – June 2012

| Medication | United Healthcare | MarketScan | Total |
|------------|-------------------|------------|--------|
| Dabigatran | 4,150 | 20,000 | 24,150 |
| Warfarin | 7,720 | 40,000 | 47,720 |

#### **7.6 BIAS**

Various design and analysis methods will be implemented to reduce the potential for bias in the study. We will employ new-user cohorts of NOAC medications and warfarin in order to address differences that might arise in the comparison of newer and older treatments, such as survivor bias and attrition of susceptibles. The comparator cohort will be formed from warfarin initiators with similar clinical profiles to dabigatran and other NOAC medications initiators to reduce confounding by indication. We will employ propensity score matching of NOAC/dabigatran and warfarin cohorts in order to improve the balance of the cohorts with respect to numerous variables and will further assess the balance across the matched cohorts on the basis of disease risk scores for the primary outcomes. We will use established

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

algorithms for outcome identification and only outcomes expected to be ascertained well in insurance claims.

#### 7.7 STUDY SIZE

The ability of this research program to detect a given risk increase depends on the incidence of the outcome as well as the number of cohort entrants and duration of follow-up. The study size will depend on the number of dabigatran (or other NOAC medications) and warfarin initiators who meet the study inclusion and exclusion criteria and are successfully matched into cohorts. On the basis of the outcome incidence rate observed in the comparison group in the pilot phase of this project (Phase 1) and the cumulative person-time of observation over the study period, we estimated the minimum relative rate that can be detected with 80% power for dabigatran-warfarin comparison.. During the period October 2010 – June 2012, among patients with a minimum of 12 months baseline history, no prior use of any anticoagulants, and a diagnosis of non-valvular atrial fibrillation, there are 4,158 dabigatran incident users in the UnitedHealth database and approximately 20,000 dabigatran users in MarketScan database. These dabigatran users will be matched to a similar number of warfarin incident users. Assuming that approximately 70% or patients will be matched, an average follow-up of 5 months (both based on the preliminary results from Phase 1 of the Pradaxa project) and the additional users who initiated dabigatran during July-December 2012 period, there should be slightly more 10,000 person-years of dabigatran follow-up for the initial analysis. As this project expands in 6 month increments, the persontime, along with outcomes and the ability to detect a particular relative risk will increase.

The table below provides estimates of the minimum relative rates that can be detected with 80% power for the major study outcomes under specific assumptions regarding their incidence in the comparator group (labeled "base rate") and the accrual of person-time. The base case incidence rates are the rates observed in warfarin initiators who were calendar quarter- and PS- matched to dabigatran initiators during the October 2010-June 2012 period in the UnitedHealth database (Phase 1 of the project). We conservatively assumed that the number of patients initiating dabigatran each month during July 2012 – December 2015 is equal to the average monthly number of initiators during the first half of 2012, that at least 2/3 of these patients are matched 1:1 to comparator patients, and that each patient contributes 0.41 years of follow-up time.

Table 8 Projected minimum detectable relative rates\* by reporting period

| | Phase 1<br>(NOAC<br>Cohort) | Interim<br>report 1 | Interim report 2 | Interim report 3 | Interim report 4 | Interim report 5 | Interim report 6 | Final report |
|---|---|---|---|---|---|---|---|---|
| Report Date | | Apr,<br>2014 | Jul,<br>2014 | Nov,<br>2014 | Mar,<br>2015 | Sep,<br>2015 | Mar,<br>2016 | Dec,<br>2016 |

Table 8 (con't) Projected minimum detectable relative rates\* by reporting period

| Data through<br>(MarketScan/<br>United) | Jun,<br>2012 | Dec,<br>2012 | Jun,<br>2013 | Sep/Dec,<br>2013 | Dec<br>2013/Jun<br>, 2014 | Sept/Dec,<br>2014 | Dec<br>2014/Jun<br>, 2015 | Dec,<br>2015 |
|---|---|---|---|---|---|---|---|---|
| Estimated number of matched patients | | 24,000 | 30,000 | 36,000 | 42,000 | 48,000 | 54,000 | 60,000 |
| Cumulative person-time of observation | | 10,000 | 12,350 | 14,700 | 17,050 | 19,400 | 21,750 | 24,100 |
| Outcome | Base rate † | | Minimum detectable relative rate | | | | | |
| Stroke | 31.59 | 1.24 | 1.21 | 1.19 | 1.18 | 1.17 | 1.16 | 1.15 |
| Major<br>Hemorrhage | 66.72 | 1.16 | 1.14 | 1.13 | 1.12 | 1.11 | 1.11 | 1.10 |
| Ischemic<br>stroke | 32.71 | 1.23 | 1.21 | 1.19 | 1.17 | 1.16 | 1.15 | 1.15 |
| Hemorrhagic stroke | 2.09 | 1.87 | 1.77 | 1.70 | 1.64 | 1.60 | 1.56 | 1.53 |
| MI | 14.73 | 1.35 | 1.32 | 1.29 | 1.27 | 1.25 | 1.23 | 1.22 |
| Major GI<br>bleeding | 31.63 | 1.24 | 1.21 | 1.19 | 1.18 | 1.17 | 1.16 | 1.15 |
| Hepatotoxici<br>ty | 4.20 | 1.70 | 1.62 | 1.57 | 1.52 | 1.49 | 1.46 | 1.43 |

<sup>\*</sup> This table reports the minimum relative rate that can be detected with 80% power assuming an alpha level of 0.05 and a 2-sided test.

<sup>†</sup> Base rate is incidence rate per 1,000 Person-Years observed in warfarin initiators matched to dabigatran during the October 2010-June 2012 period in the UnitedHealth database

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7.9 DATA ANALYSIS

All analysis will be performed with SAS Inc, Version 9.3.

#### 7.9.1 MAIN ANALYSIS

All analyses will be conducted in both data sources and may be combined in pooled analyses if appropriate, based on homogeneity of treatment effect. Pooling of results across data sources will correspond to a weighted average effect (as in a fixed effects meta-analysis) using the Mantel-Haenszel method. [R97-0509] Heterogeneity will be assessed by comparing the treatment effect point estimates across data sources. If there is a difference >30% in the overall effect measure for a primary outcome across the two data sources, we will conduct an additional investigation that assesses treatment effect within levels of protocol-specified subgroups (Section 6.9.2) separately by a database. If treatment effect is different across levels of the subgroup variable within a data source, and the distribution of this subgroup variable differs by data source, then the pooling will be conducted within strata of the subgroup variable or variables across which heterogeneity is observed to account for this heterogeneity (see Section 6.2 for more details). In each data source, we will compare distributions of socio-demographic, clinical and utilization characteristics among initiators of different anticoagulant agents, and calculate event rates during follow-up for each of the specified outcomes.

Unadjusted and adjusted relative risks (hazard ratios) and rate differences will be estimated. In adjusted analyses, we will use propensity score (PS) matching to balance potential confounders. [R13-1120] [R12-1912] PS will be derived from predicted probabilities of treatment initiation, given all measured covariates. We will estimate the primary propensity score for each patient using a logistic regression model that includes all pre-defined covariates (from Section 6.4.3). The propensity score will be used to match dabigatran initiators to initiators of warfarin on a 1:1 fixed ratio basis using a nearest-neighbor algorithm and a caliper of 0.05. In addition, patients will be matched on calendar quarter of initiation. Individual covariates will be further tabulated and compared across matched cohorts. If substantial covariate imbalance between dabigatran and warfarin is noted as assessed by a standardized difference >0.1, then we will further adjust the outcome models for HAS-BLED and CHA<sub>2</sub>DS<sub>2</sub>-VASc score as Cohort Phase 1 results indicated that these scores include all the variables typically imbalanced.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

We will plot post-PS-matching Kaplan-Meier curves for event-free survival as a function of the duration of use of the index anticoagulant agent to evaluate the proportionality of hazards.

Proprietary confidential information  $\odot$  2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The secondary analyses will involve other NOAC medications as compared to warfarin. Other NOACs will include rivaroxaban, apixaban and others once they become available for stroke prevention in NVAF patients. We will monitor the number of patients initiating other NOACs and provide these numbers along with power calculations for primary outcomes at each interim report. Once sufficient numbers have accrued, and sufficient follow up time is available, these other NOAC initiators will be separately matched to warfarin initiators and primary analyses (and further/sensitivity analyses if numbers allow) as described above for dabigatran-warfarin comparison will be done.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.10 QUALITY CONTROL

All aspects of data analysis will be conducted according to standard procedures of the Division of Pharmacoepidemiology. Programming for this project will be conducted by a primary analyst and validated by a separate analyst (validation analyst). For all data processing and analysis steps, the validation analyst will review the program along with input and output data sets, and for select steps of the project will employ double programming techniques to reduce the potential for programming errors.

#### 7.11 LIMITATIONS OF THE RESEARCH METHODS

As an observational study, there are inherent limitations with respect to potential for alternate explanations for any observed association.

The source claims data include limitations with respect to certainty of capture of exposure, covariates, and outcomes. As a comprehensive insurance database, essentially all billable medical services will result in claims for reimbursement, so that certainty of capture is tied to likelihood of a claim being submitted to the insurer.

Given the characteristics of the UnitedHealth data (commercial health insurer), patients older than 65 years will be under-represented in the data. Only approximately 35% of incident dabigatran users during the 2010-2011 period were 65 years of age and older. As NVAF also predominately affects older population, it will be under-represented in the data as well.

Although duration of atrial fibrillation may represent a risk factor for study outcomes, this covariate will be incompletely captured since the patient history in the dataset is relatively short (at least 6 months, and an average of approximately 2 years), and a first claim within the database may not represent atrial fibrillation onset since the condition is typically not diagnosed at its onset.

Dosing of warfarin in clinical practice is complicated, and estimating dose and duration of exposure based on healthcare utilization data is therefore challenging. The "days' supply" field is expected to be most meaningful, but the potential for misclassification exists.

There are a number of covariates, such as the type of atrial fibrillation, cause-specific mortality, BMI, smoking, that are not directly assessed in a health insurer database. Information on formulary and reimbursement is not available for MarketScan data. Further, some covariates that can be directly assessed through diagnosis and procedure codes (such as renal dysfunction) have uncertain sensitivity, specificity, and predictive value. Estimation of creatinine clearance even in the subgroup of patients with laboratory values present is not feasible as information on height and weight is not available. A modified MDRD equation is going to be used (see Further Analysis section), which - although found to accurately estimate GFR from serum creatinine measurements - is not used for dosing. In our study, however, we will only use it to assess balance between exposure cohorts.

In addition, medication use in United Healthcare data and MarketScan data - as in all administrative healthcare databases - is restricted to prescription drug medication.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Consequently, the use of over-the-counter (OTC) medications (e.g., OTC aspirin) is not captured. In addition, exposure is assessed based on prescription pick-up at a pharmacy and might be misclassified in "as treated" analysis if patients do not take their medications. However, misclassification of prescription drug exposure is generally considered less than in other exposure assessment approaches, including physician prescribing records and patient self-reporting. [P13-03077] [P13-03078]

## 7.12 OTHER ASPECTS

Any other aspect of the research method not covered by the previous sections.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. PROTECTION OF HUMAN SUBJECTS

Data analysis personnel will have access to patients protected health information (PHI) while linking databases and constructing study variables. After data linkage and variable construction is completed, the subjects' PHI will be deleted from the study database, therefore posing minimal risk to patients' privacy.

This study will be submitted to the Institutional Review Board (IRB) of the

.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 9. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This will be a retrospective observational study; all patient data will be de-identified and analyzed in aggregate. Individual patient safety related information will not be captured during this study. Thus, individual safety reporting is not applicable for this study.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The interim and final reports will consist of a description of the methods, including patient selection and variable definitions along with tabular summaries of cohort characteristics, numbers of patients receiving each anticoagulant and associated follow-up time. Counts of outcomes and corresponding rates and measures of association will be presented. The tabular results will be followed by an interpretive summary along with a discussion of the findings and implications.

The scheduling of communication of interim results will be specified in a separate document.

Manuscripts describing this work will be submitted for publication in peer-review journals. Findings may also be submitted for presentation at scientific conferences.

## 11. REFERENCES

- P06-10925 Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ. Validation of clinical classification schemes for predicting stroke: results from the National Registry of Atrial Fibrillation. JAMA 2001;285:2864-70.
- P08-02098 Myers RP, Leung Y, Shaheen AA, Li B. Validation of ICD-9-CM/ICD-10 coding algorithms for the identification of patients with acetaminophen overdose and hepatotoxicity using administrative data. BMC Health Serv Res 2007;7:159.
- P09-11669 Connolly SJ, Ezekowitz MD, Yusuf S, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med 2009;361:1139-51.
- P11-11875 Potpara TS, Lip GY. New anticoagulation drugs for atrial fibrillation. Clin Pharmacol Ther 2011;90:502-6.
- P12-01676 You JJ, Singer DE, Howard PA, et al. Antithrombotic therapy for atrial fibrillation: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest 2012;141:e531S-75S.
- P12-05791 FDA draft guidance for industry on Drug Interaction Studies Study Design, Data Analysis, and Implications for Dosing and Labelling. Feb 2012. at website: fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM292362.pdf.)
- P12-08895 Rassen JA, Glynn RJ, Rothman KJ, Setoguchi S, Schneeweiss S. Applying propensity scores estimated in a full cohort to adjust for confounding in subgroup analyses. Pharmacoepidemiol Drug Saf 2012;21:697-709.
- P12-11192 Camm AJ, Lip GY, De Caterina R, et al. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: An update of the 2010 ESC Guidelines for the management of atrial fibrillation \* Developed with the special contribution of the European Heart Rhythm Association. Europace 2012;14:1385-413.
- P13-03077 West SL, Strom BL, Freundlich B, Normand E, Koch G, Savitz DA. Completeness of prescription recording in outpatient medical records from a health maintenance organization. J Clin Epidemiol 1994;47:165-71.
- P13-03078 West SL, Savitz DA, Koch G, Strom BL, Guess HA, Hartzema A. Recall accuracy for prescription medications: self-report compared with database information. Am J Epidemiol 1995;142:1103-12.
- R03-1232 Go AS, Hylek EM, Borowsky LH, Phillips KA, Selby JV, Singer DE. Warfarin use among ambulatory patients with nonvalvular atrial

| | fibrillation: the anticoagulation and risk factors in atrial fibrillation (ATRIA) study. Ann Intern Med 1999;131:927-34. |
|---|---|
| R05-0358 | Cushman M, Tsai AW, White RH, et al. Deep vein thrombosis and pulmonary embolism in two cohorts: the longitudinal investigation of thromboembolism etiology. Am J Med 2004;117:19-25. |
| R10-5332 | Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest 2010;137:263-72. |
| R10-6394 | Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest 2010;138:1093-100. |
| R11-2274 | Cunningham A, Stein CM, Chung CP, Daugherty JR, Smalley WE, Ray WA. An automated database case definition for serious bleeding related to oral anticoagulant use. Pharmacoepidemiol Drug Saf 2011;20:560-6. |
| R11-4190 | Granger CB, Alexander JH, McMurray JJ, et al. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med 2011;365:981-92. |
| R11-4223 | Patel MR, Mahaffey KW, Garg J, et al. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med 2011;365:883-91. |
| R11-4316 | Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of Medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. Am Heart J 2004;148:99-104. |
| R11-4329 | Winkelmayer WC, Schneeweiss S, Mogun H, Patrick AR, Avorn J, Solomon DH. Identification of individuals with CKD from Medicare claims data: a validation study. Am J Kidney Dis 2005;46:225-32. |
| R11-4334 | Birman-Deych E, Waterman AD, Yan Y, Nilasena DS, Radford MJ, Gage BF. Accuracy of ICD-9-CM codes for identifying cardiovascular and stroke risk factors. Med Care 2005;43:480-5. |
| R11-4887 | Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. Pharmacoepidemiol Drug Saf 2010;19:596-603. |
| R12-0541 | Friberg L, Rosenqvist M, Lip GY. Evaluation of risk stratification schemes for ischaemic stroke and bleeding in 182 678 patients with atrial fibrillation: the Swedish Atrial Fibrillation cohort study. Eur Heart J 2012;33:1500-10. |
| R12-1912 | Rosenbaum PR, Rubin DB. The central rol of the propensity score in observational studies for causal effects. Biometrica 1983:41-55. |

| R12-1912 | Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. Biometrica 1983:41-55. |
|---|---|
| R13-0519 | Benesch C, Witter DM, Jr., Wilder AL, Duncan PW, Samsa GP, Matchar DB. Inaccuracy of the International Classification of Diseases (ICD-9-CM) in identifying the diagnosis of ischemic cerebrovascular disease. Neurology 1997;49:660-4. |
| R13-0520 | Kokotailo RA, Hill MD. Coding of stroke and stroke risk factors using international classification of diseases, revisions 9 and 10. Stroke 2005;36:1776-81. |
| R13-0521 | Molnar AO, Coca SG, Devereaux PJ, et al. Statin use associates with a lower incidence of acute kidney injury after major elective surgery. J Am Soc Nephrol 2011;22:939-46. |
| R13-0522 | Tamariz L, Harkins T, Nair V. A systematic review of validated methods for identifying venous thromboembolism using administrative and claims data. Pharmacoepidemiol Drug Saf 2012;21 Suppl 1:154-62. |
| R13-0523 | Glynn RJ, Gagne JJ, Schneeweiss S. Role of disease risk scores in comparative effectiveness research with emerging therapies. Pharmacoepidemiol Drug Saf 2012;21 Suppl 2:138-47. |
| R13-0524 | Hansen B. The prognostic analogue of the propensity score. Biometrika 2008;95:481-8. |
| R13-0525 | Schneeweiss S, Rassen JA, Glynn RJ, Avorn J, Mogun H, Brookhart MA. High-dimensional propensity score adjustment in studies of treatment effects using health care claims data. Epidemiology 2009;20:512-22. |
| R13-0526 | Huybrechts KF, Rothman KJ, Silliman RA, Brookhart MA, Schneeweiss S. Risk of death and hospital admission for major medical events after initiation of psychotropic medications in older adults admitted to nursing homes. CMAJ 2011;183:E411-9. |
| R13-0527 | Rassen JA, Schneeweiss S. Using high-dimensional propensity scores to automate confounding control in a distributed medical product safety surveillance system. Pharmacoepidemiol Drug Saf 2012;21 Suppl 1:41-9. |
| R13-0528 | Patorno E, Bohn RL, Wahl PM, et al. Anticonvulsant medications and the risk of suicide, attempted suicide, or violent death. JAMA 2010;303:1401-9. |
| R13-0540 | Rule AD, Larson TS, Bergstralh EJ, Slezak JM, Jacobsen SJ, Cosio FG. Using serum creatinine to estimate glomerular filtration rate: accuracy in good health and in chronic kidney disease. Ann Intern Med 2004;141:929-37. |
| R13-1120 | Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. Pharmacoepidemiol Drug Saf 2010;19:858-68. |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| R13-4176 | Olesen JB, Lip GY, Hansen PR, et al. Bleeding risk in 'real world' patients with atrial fibrillation: comparison of two established bleeding prediction schemes in a nationwide cohort. J Thromb Haemost 2011;9:1460-7. |
|---|---|
| R13-5082 | Giugliano RP, Ruff CT, Braunwald E, et al. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med 2013;369:2093-104. |
| R14-0052 | Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiol Drug Saf 2012;21 Suppl 1:100-28. |
| R96-0690 | Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41. |
| R97-0509 | Mantel N, Haenszel W. Statistical aspects of the analysis of data from retrospective studies of disease. Journal of the National Cancer Institute 1959;22:719-48. |

# 12. FUNDING

Boehringer Ingelheim GmbH

# 13. ANNEX

## **ANNEX 1: LIST OF STAND-ALONE DOCUMENTS**

None

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Table A3 Follow-up and outcomes among matched cohorts

| Group | Size | Follow-up (P-Y) | Outcome events | Incidence Rate | HR | 95% CI |
|---|---|---|---|---|---|---|
| Dabigatran | N | | | | | |
| Warfarin | N | | | | | |

This table will be repeated for each of the outcomes

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Table A4 Follow-up and distribution of reasons for discontinuation

| | | Follow-up (years) | | Reasons for discontinuation (N, %) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | Size | Mean | Median | Max | Discon<br>tinue | Switch | Event | Disenro<br>Ilment | Death | Nursing<br>home<br>admission |
| Dabigatran | N | | | | | | | | | |
| Warfarin | N | | | | | | | | | |

This table will be repeated for each of the outcomes.

## Boehringer Ingelheim Protocol for observational studies based on existing data 1160.207


c02336230-01

### **ANNEX 4 STUDY FIGURES**



NOAC: New Oral Anticoagulant

Figure A1 Patient Selection Flow Diagram (CONSORT Style)

This figure will be produced for each interim report and the final report

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Figure A2 Survival curves (time to event)

Separate figures to be created for each of the study outcomes. These figures will be produced for each interim report and the final report and displayed in the respective report.



### APPROVAL / SIGNATURE PAGE

**Document Number:** c02336230 **Version Number:** 1.0

**Document Name:** 1160-0207-protocol

Title: Sequential Expansion of Comparative Effectiveness of Oral Anticoagulants: A Cohort

Study

## **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | <b>Date Signed</b> |
|---|---|---|
| Approval-EU Qualified Person<br>Pharmacovigilance | | 25 Feb 2014 15:48 CET |
| Approval-Pharmacovigilance<br>Representative | | 25 Feb 2014 16:24 CET |
| Author-Other | | 25 Feb 2014 17:11 CET |
| Approval- Pharmacovigilance | | 25 Feb 2014 17:38 CET |
| Approval-Other | | 27 Feb 2014 11:41 CET |
| Approval-Team Member Medical<br>Affairs | | 28 Feb 2014 11:03 CET |
| Verification-Paper Signature<br>Completion | | 28 Feb 2014 19:04 CET |
| Approval-Therapeutic Area | | 05 Mar 2014 13:21 CET |

Boehringer IngelheimPage 2 of 2Document Number: c02336230Version Number: 1.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by | Date Signed |
|--------------------------------|-------------|
|--------------------------------|-------------|